CLINICAL TRIAL: NCT04734769
Title: Embryos With Preimplantation Genetic Testing for Aneuploidies (PGT-A) Inconclusive Result: Clinical Implications
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: IVI Vigo (Other)
Collaborators: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other); Juno Therapeutics, Inc., a Bristol-Myers Squibb Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 2011-VGO-095-EM
Record Dates: First submitted 2021-01-27; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Embryo Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cycles of embryo transfer from patients with at least one euploid embryo (no rebiopsy group): Collect retrospectively clinical data on reproductive outcomes
  Interventions: Other: Collect retrospectively clinical data on reproductive outcomes
- Rebiopsy group:: Collect retrospectively clinical data on reproductive outcomes
  Interventions: Other: Collect retrospectively clinical data on reproductive outcomes

INTERVENTIONS:
Other: Collect retrospectively clinical data on reproductive outcomes — Collect retrospectively clinical data on reproductive outcomes

SUMMARY:
One of the most remarkable improvements in trophoectoderm cells biopsy is the robustness of diagnosis as result of analyzing multiple cells. However, there is a proportion of embryos that lack of diagnosis due to amplification failure or inconclusive results ranging between 0,4% and 6%. Information about embryo repeated biopsy after an inconclusive result in a first biopsy is very scarce. No specific conclusions can be drawn, due to the limited information currently available concerning reproductive outcomes for patients who had embryo transfer after a second biopsy, due to a first one having an inconclusive result. Investigators purpose a multicenter retrospective observational study with the aim to evaluate the reproductive potential of re-biopsied blastocyst with inconclusive results on preimplantation genetic screening for aneuploidy (PGT-A) using the implantation rate (IR) and ongoing pregnancy rate (OPR) as principal variables.

DETAILED DESCRIPTION:
The main objective of assisted reproduction technologies (ART) is to achieve a healthy live newborn. The selection of an euploid embryo using PGT-A, offers theoretical advantages including increased implantation rate, reduced abortion rate, and reduces the time to achieve an ongoing pregnancy.

Certain advances in ART such as vitrification or improvement in culture media makes safer the PGT-A procedure. As a result of these improvements, embryo biopsy has been driven from blastomere to trophectoderm biopsy at blastocyst stage for preimplantional genetic testing for aneuploidy analysis (PGT-A 2.0) and it is now the method of choice for PGT-A in many centers. Trophectoderm biopsy presents advantages over the use of blastomere biopsy: 1. It allows obtaining around 6-10 cells without reducing the potential for pre-embryo development or its ability to implant. 2. Greater strength in the results, since it reduces false diagnoses associated with factors such as mosaicism. 3. It allows a combined study for monogenic mutations, aneuploidy screening and / or structural alterations.

The frequency of inconclusive results in PGT-A varies depending on the embryonic stage used, with values of 9-10% of the total embryos analyzed for single blastomere biopsy and between 2-6% when trophectoderm cells are biopsied.

These inconclusive results, mainly in couples without euploid embryos available to transfer, cause them uncertainty and disappointment. In these situations, it is advisable to guide patients in making decisions about what to do with these pre-embryos through genetic counselling. Patients must decide if they wish to reject them, to transfer them without the certainty of a reliable diagnosis or to re-analyze them. Scientific literature reporting these types of inconclusive results and that give advice about its possible etiology are scarce. There is no clear evidence about the impact of double biopsy, double vitrification-warming or if transferring embryos with inconclusive results, is safe for achieving a healthy newborn. The objective of this review is to learn from the published studies about the safety of embryo re-analysis and its potential reproductive outcome when there are embryos with inconclusive results after PGT, in order to offer adequate counselling for patients.

ELIGIBILITY:
Inclusion Criteria:

* Cycles of embryo transfer from patients with at least one euploid embryo (no rebiopsy group):
* Women age 18-45 years.
* PGT-A Indication.
* All embryos with informative results.
* Women age 18-45 years.
* PGT-A Indication.
* At least one embryo result with lack of diagnosis.
* At least one rebiopsied embryo.
* At least one euploid result from rebiopsied embryo.
* Single embryo transfer.

Exclusion Criteria:

Double embryo transfer

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: All patients with indication of PGT-A (advanced maternal age, male factor, recurrent pregnancy loss, recurrent implantation failure, previous aneuploidy pregnancy) with differed single embryo transfer.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-02-20 (Estimated); Primary Completion 2021-02-21 (Estimated); Study Completion 2022-11-25 (Estimated)

PRIMARY OUTCOMES:
Implantation rate | Since July 2019 to December 2020
  Analyze implantation rate in the groups

CONTACTS AND LOCATIONS:
Overall Officials: Elkin Muñoz, Study Director — IVI Vigo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cobo A, Castello D, Vallejo B, Albert C, de los Santos JM, Remohi J. Outcome of cryotransfer of embryos developed from vitrified oocytes: double vitrification has no impact on delivery rates. Fertil Steril. 2013 May;99(6):1623-30. doi: 10.1016/j.fertnstert.2013.01.106. Epub 2013 Feb 14. PMID 23415972
- [Background] Chen HH, Huang CC, Cheng EH, Lee TH, Chien LF, Lee MS. Optimal timing of blastocyst vitrification after trophectoderm biopsy for preimplantation genetic screening. PLoS One. 2017 Oct 5;12(10):e0185747. doi: 10.1371/journal.pone.0185747. eCollection 2017. PMID 28982142